CLINICAL TRIAL: NCT06353633
Title: The Effect of Exclusion Diet for Crohn's Disease Plus Enteral Nutrition on Children and Adolescents With Crohn's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: AHekmatdoost
Record Dates: First submitted 2024-02-23; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Inflammatory Bowel Diseases
Keywords: PEN
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Food, Formulated; Elimination Diets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exclusion diet along with formula (Active Comparator)
  Interventions: Dietary Supplement: formula; Behavioral: exclusion diet
- A group that receives only exclusion diet (Active Comparator)
  Interventions: Behavioral: exclusion diet

INTERVENTIONS:
Dietary Supplement: formula — The calories needed by the person are calculated and half of the calories are provided by formulas and the other half based on the elimination diet
  Arms: exclusion diet along with formula
Behavioral: exclusion diet — In this group, only the elimination diet is considered as an intervention

SUMMARY:
In this study, children and adolescents with active Crohn's disease are placed in two intervention groups, the first group receives only an exclusion diet and the second group receives an exclusion diet plus formula.

ELIGIBILITY:
Inclusion Criteria:

* children aged 4 to 18 years with active Crohn's disease
* Pediatric Crohn's Disease Activity Index (PCDAI) ≥10 and ≤40

Exclusion Criteria:

* Patients who receiving concurrent remission-inducing drugs such as steroids, 5-ASA, methotrexate, or antibiotics, as well as patients receiving induction doses of a biologic

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-04-10 (Estimated); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
PCDAI | 8 weeks
  pediatric chron disease activity index
CRP | 8 weeks
  c-reactive protein
ESR | 8 weeks
  erythrocyte sedimentation rate
FC | 8 weeks
  fecal calprotectin
Alb | 8 weeks
  serum albumin

SECONDARY OUTCOMES:
Arm Circumferance | 8 weeks
  the circumference of the arm
BMI | 8 weeks
  body mass index
Height | 8 weeks
  height measurement
weight | 8 weeks
  body weight

CONTACTS AND LOCATIONS:
Overall Officials: Azita Hekmatdoost, MD, PhD, Study Director — NNFTRI

IPD SHARING:
Plan to Share IPD: Undecided